CLINICAL TRIAL: NCT07095725
Title: Effect of Primary Dysmenorrhea on Abdominal and Back Muscles Activity in Young Adult Females
Brief Title: Effect of Primary Dysmenorrhea on Muscle Activity in Young Adult Females
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahenour Esmail Taha, Teaching Assistant, Cairo University
Other Study IDs: P.T.REC\012\005884
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Primary Dysmenorrhea
Keywords: Muscle Activity; Maximum Voluntary Contraction; EMG; Primary Dysmenorrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Mild dysmenorrhea: Females with mild PD, scoring (1-4) on the WaLLID scale.
  Interventions: Diagnostic Test: Record EMG maximum amplitude from rectus abdominis, erector spinae L3 level
- Group B: Moderate dysmenorrhea: Females with moderate PD, scoring (5-7) on the WaLLID scale.
  Interventions: Diagnostic Test: Record EMG maximum amplitude from rectus abdominis, erector spinae L3 level
- Group C: Severe dysmenorhhea: Females with severe PD, scoring (8-12) on the WaLLID scale.
  Interventions: Diagnostic Test: Record EMG maximum amplitude from rectus abdominis, erector spinae L3 level

INTERVENTIONS:
Diagnostic Test: Record EMG maximum amplitude from rectus abdominis, erector spinae L3 level — EMG Electrode Placement and Muscle Assessment:
  Electrodes for the rectus abdominis were placed longitudinally at the umbilical level. For the erector spinae, L3 was located using a line between the posterior superior iliac crests, and electrodes were placed ~3 cm lateral to the L3 spinous process.
  Assessment:
  Rectus Abdominis: In the crook-lying position, participants performed a slow curl-up (~35-40°), holding for 10 seconds.
  Erector Spinae: In the prone position with a 10-cm pad under the abdomen, participants lifted the upper body with neutral cervical alignment for 10 seconds.
  Each test was repeated three times with 2-minute rest intervals.

SUMMARY:
This study aims to investigate the effect of primary dysmenorrhea on the activity of the abdominal and back muscles in young adult females.

DETAILED DESCRIPTION:
PD is highly prevalent in females, which directly influences their quality of life, physical function and performance. A study conducted in Palestine has shown that over half of university students with dysmenorrhea tend to skip university lectures due to painful menses.

PD is commonly associated with visceral pain and various musculoskeletal symptoms, including abdominal and back pain (Yacubovich et al., 2019). This can reduce the maximum voluntary contraction of the affected muscles, compromising their ability to provide adequate support and stability (Merkle et al., 2020). Persistent pain can disrupt postural stability and balance, raising the risk of injury by compromising stability and muscle function.

Research highlights the impact of primary dysmenorrhea (PD) on muscle function, particularly in the abdominal and back muscles, contributing to pain and reduced stability. Oladosu et al. (2018) found that abdominal muscle activity precedes menstrual pain, suggesting a neuromuscular link. Similarly, Karakus et al. (2022) and Álvarez et al. (2024) reported altered activation and reduced endurance in stabilizing muscles, including the transversus abdominis, obliques, and lumbar multifidus, with muscle thinning that may impair spinal stability. These studies emphasize PD's effect on muscle function, but further research is needed to explore variations across severities and guide effective treatments.

When these weakened muscles because of dysmenorrhea are subjected to increased or sudden activity during daily living tasks, such as lifting, bending, or other physical exertions, the risk of injury to the structures they are designed to protect is significantly heightened (Escamilla et al., 2010; Polat et al., 2022).

However, to the best of the authors' knowledge, no research has yet explored the relationship of abdominal and back muscle activity patterns to PD and their variations across different severities of dysmenorrhea, which directly contributes to females' quality of life.

Understanding this association could have significant clinical implications and contribute to new knowledge that helps physical therapists determine the need for custom-designed prevention and treatment programs for females with PD. By raising awareness of the potential musculoskeletal risks associated with PD, this study emphasizes the importance of minimizing strenuous activities during menstruation to reduce muscle strain or injury, ultimately enhancing overall health and well-being during this period.

ELIGIBILITY:
Inclusion Criteria:

* All females clinically diagnosed with PD, as confirmed and referred by a gynecologist.
* Age ranges from 18 to 25 years.
* BMI ranges from 20 to 25 kg/m2 .
* Onset of menstrual pain 6-24 months after menarche.
* Having a regular menstrual cycle (28 ± 7 days with no intermittent bleeding).
* Their PD symptoms will be determined according to the WaLLID questionnaire and will be classified into mild PD (1-4), moderate PD (5-7), severe PD (8-12).
* All participants are virgins.

Exclusion Criteria:

* Menstrual irregularity.
* Use of antidepressant or steroid drugs.
* Secondary dysmenorrhea.
* Musculoskeletal problems in the abdominal region, pelvic region, or spine.
* Surgical history involving the abdominal region, pelvic region, or spine in the last year.
* Any psychiatric or gynecological problems.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Young females with primary dysmenorrhea
Study Population: Young adult females with primary dysmenorrhea
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Activity of rectus abdominis muscle | 3 months
  Maximum voluntary contraction in (μV) of rectus abdominis using electromyography device (EMG)
Activity of erector spinae muscle at L3 vertebrae Level | 3 Month
  Maximum voluntary contraction in (μV) of erector spinae at L3 Level using electromyography device (EMG)

CONTACTS AND LOCATIONS:
Overall Officials: Mahenour Esmail Shendy, Bachelor of Physical Therapy, Principal Investigator — Teaching Assistant of Physical Therapy For Women's Health- Misr University for Science and Technology; Doaa Ahmed Osman, Assistant Professor, Study Chair — Physical Therapy for Women's Health - Faculty of Physical Therapy- Cairo University; Manal Ahmed Elshafei, Lecturer, Study Director — Physical Therapy for Women's Health - Faculty of Physical Therapy- Cairo University; Ihab Kamal Younis, lecturer, Study Director — Obstetrics and Gynecology department - Faculty of Medicine Misr university for science and technology
Locations (1):
- Misr University for Science and Technology, Giza, Egypt